CLINICAL TRIAL: NCT07148687
Title: Effect of ChatGPT and DeepSeek-Guided Rehabilitation on Clinical Outcomes in Individuals With Subacromial Pain Syndrome
Brief Title: ChatGPT and DeepSeek-Assisted Rehabilitation in Subacromial Pain
Acronym: LLM-RehabSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Omer Alperen Gurses, PhD, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025/874
Record Dates: First submitted 2025-08-03; First posted 2025-08-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Subacromial Pain Syndrome
Keywords: ChatGPT; DeepSeek; Large Language Models; Shoulder Rehabilitation; Subacromial Pain; Artificial Intelligence

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to three parallel groups:
  1. standard physiotherapy combined with a conventional exercise program for subacromial pain syndrome based on current clinical guidelines,
  2. standard physiotherapy combined with ChatGPT-guided exercises, and
  3. standard physiotherapy combined with DeepSeek-guided exercises.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants were informed that they would receive one of several supervised exercise-based rehabilitation programmes for subacromial pain syndrome, but were not informed of their specific group assignment or the use of large language models. The physician establishing the diagnosis and the physiotherapist performing all outcome assessments are blinded to group allocation. Treating physiotherapists are aware of group assignment but are not involved in outcome assessments or data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Exercise Group (Active Comparator): Participants receive standard physiotherapy combined with a conventional exercise program for subacromial pain syndrome based on evidence-based clinical guidelines. Each group included 23 participants who completed the 6-week intervention and were included in the final analysis.
  Interventions: Behavioral: Conventional Exercise Program
- ChatGPT-Guided Exercise Group (Experimental): Participants receive standard physiotherapy combined with a conventional exercise program for subacromial pain syndrome based on evidence-based clinical guidelines. Each group included 23 participants who completed the 6-week intervention and were included in the final analysis.
  Interventions: Behavioral: ChatGPT-Guided Rehabilitation
- DeepSeek-Guided Exercise Group (Experimental): Participants receive standard physiotherapy combined with exercises generated by the DeepSeek-R1 large language model. Each group included 23 participants who completed the 6-week intervention and were included in the final analysis.
  Interventions: Behavioral: DeepSeek-Guided Rehabilitation

INTERVENTIONS:
Behavioral: Conventional Exercise Program — Exercise protocol targeting subacromial pain syndrome, including shoulder mobility, strengthening, and posture correction exercises based on established clinical guidelines.
  Arms: Standard Exercise Group
Behavioral: ChatGPT-Guided Rehabilitation — AI-generated exercise recommendations from ChatGPT-4 tailored to the patient's profile and applied under physiotherapist supervision.
  Arms: ChatGPT-Guided Exercise Group
Behavioral: DeepSeek-Guided Rehabilitation — Personalized rehabilitation exercises generated by DeepSeek-R1 and implemented under physiotherapist guidance.
  Arms: DeepSeek-Guided Exercise Group

SUMMARY:
This study aims to evaluate the effects of rehabilitation programs supported by artificial intelligence-based large language models (LLMs), specifically ChatGPT and DeepSeek, in individuals with subacromial pain syndrome (SAPS). Participants will be randomly assigned to one of three groups: standard physiotherapy, standard physiotherapy plus ChatGPT-guided exercises, and standard physiotherapy plus DeepSeek-guided exercises. Outcomes including pain, disability, quality of life, muscle strength, and joint range of motion will be assessed before and after a 6-week intervention. The results will help determine whether AI-generated exercise recommendations can enhance clinical outcomes when combined with conventional physiotherapy.

DETAILED DESCRIPTION:
This completed randomized controlled trial investigated the clinical effects of integrating AI-generated exercise recommendations into conventional physiotherapy for individuals with subacromial pain syndrome (SAPS). A total of 82 individuals were assessed for eligibility; 7 were excluded for not meeting inclusion criteria. Seventy-five participants provided consent and were randomized equally to 3 groups (n=25 each): (1) conventional physiotherapy plus a conventional exercise program, (2) conventional physiotherapy plus ChatGPT-guided exercises, and (3) conventional physiotherapy plus DeepSeek-guided exercises. Interventions were delivered over 6 weeks (3 supervised sessions/week).

Six participants discontinued the intervention due to scheduling conflicts (2 per group). Sixty-nine participants completed the 6-week intervention and were included in the final analysis (n=23 per group).

Co-primary outcomes were pain intensity (NPRS: rest, activity, night), shoulder pain and disability (SPADI), and health-related quality of life (SF-12 PCS/MCS), assessed at baseline and 6 weeks. Secondary outcomes included DASH, range of motion, isometric strength (Kinvent K-Force; Newtons), kinesiophobia (TSK), pain catastrophizing (PCS), emotional status (HADS), and shoulder function (ASES, WORC).

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 65
* Having been diagnosed with Subacromial Pain Syndrome (SAPS) for at least four weeks, diagnosed through clinical and physical examination
* Actively maintaining shoulder range of motion
* Being cognitively and physically capable of participating in an exercise program
* Agreeing to participate voluntarily in the research process and providing written consent

Exclusion Criteria:

* Presence of other shoulder pathologies such as rotator cuff tear, frozen shoulder, glenohumeral instability, or labrum tear
* Presence of conditions included in the differential diagnosis such as cervical radiculopathy, neurological disorders, rheumatological diseases, or fibromyalgia
* History of shoulder surgery within the last 6 months
* Pregnancy
* History of systemic or neuromuscular disease
* Refusal to consent to voluntary participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2025-09-25 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Disability (Shoulder Pain and Disability Index, SPADI) | Baseline and after 6 weeks of intervention
  Disability related to shoulder pain will be measured.Shoulder Pain and Disability Index (0-100; higher scores indicate worse disability).

SECONDARY OUTCOMES:
Change in upper extremity function (DASH) | Baseline and after 6 weeks
  Functional status of the arm, shoulder, and hand will be assessed using the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire. Higher scores indicate greater disability.
Change in shoulder range of motion (ROM) | Baseline and after 6 weeks
  Active range of motion in shoulder flexion, extension, abduction, internal and external rotation will be measured using a standard manual goniometer.
Change in Quality of Life (Short Form-12, SF-12) | Baseline and after 6 weeks of intervention
  Health-related quality of life will be evaluated.Short Form-12 (Physical Component 12-48; Mental Component 12-48; higher scores indicate better quality of life).
Change in Pain Intensity (Numeric Pain Rating Scale, NPRS) | Baseline and after 6 weeks of intervention
  Pain intensity will be assessed using the Numeric Pain Rating Scale (NPRS) at rest, during activity, and at night. Numeric Pain Rating Scale (0-10; higher scores indicate worse pain).
Change in shoulder and elbow muscle strength (K-Force) | Baseline and after 6 weeks
  Isometric muscle strength of shoulder and elbow flexion, extension, and rotation will be assessed using the Kinvent K-Force digital dynamometer. Values will be recorded in Newtons.
Change in Kinesiophobia (Tampa Scale for Kinesiophobia, TSK) | Baseline and after 6 weeks
  Kinesiophobia will be measured using the Tampa Scale for Kinesiophobia (TSK). Tampa Scale for Kinesiophobia (17-68; higher scores indicate greater fear of movement).
Change in shoulder function (American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form, ASES) | Baseline and after 6 weeks
  Shoulder function will be evaluated using the American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form (ASES). ASES (0-100; higher scores indicate better shoulder function).
Change in Pain Catastrophizing (Pain Catastrophizing Scale, PCS) | Baseline and after 6 weeks of intervention
  Pain catastrophizing will be assessed.Pain Catastrophizing Scale (0-52; higher scores indicate worse catastrophizing).
Change in Emotional Status (Hospital Anxiety and Depression Scale, HADS) | Baseline and after 6 weeks of intervention
  Anxiety and depression will be evaluated.Hospital Anxiety and Depression Scale (0-21 for Anxiety subscale, 0-21 for Depression subscale; higher scores indicate worse symptoms).
Change in disease-specific quality of life (Western Ontario Rotator Cuff Index, WORC) | Baseline and after 6 weeks of intervention
  Disease-specific quality of life in patients with shoulder pathology will be measured.WORC (0-2100; higher scores indicate worse symptoms / lower quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University Training and Research Hospital, Physical Medicine and Rehabilitation Department, Kırşehir, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical restrictions and institutional policy. The study was not designed with external data sharing in scope.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT07148687/Prot_SAP_000.pdf